CLINICAL TRIAL: NCT03593967
Title: Project ARTISAN: Fostering Aspiration and Resilience Through Intergenerational Storytelling and Arts-based Narratives
Acronym: ARTISAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanyang Technological University (Other)
Collaborators: National Museum of Singapore (Unknown); TOUCH Community Services (Unknown); National Arts Council (Unknown); Nanyang Polytechnic (Other); NgeeAnn Polytechnic (Unknown)
Responsible Party: Principal Investigator, Andy Hau Yan Ho, PhD, EdD, Assistant Professor, Nanyang Technological University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB-2018-01-005
Record Dates: First submitted 2018-06-14; First posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Intergenerational Relations; Loneliness; Identity, Social
Keywords: wellbeing; intergenerational arts; aspiration; resilience; storytelling; art making; seniors; youth
MeSH Terms: conditions — Social Identification

STUDY DESIGN:
Intervention Model Description: Based on availability of schedule, participants will sign up for one of the 4 groups available (ie. 2 intervention groups and 2 wait-list control group). Wellbeing and self-concept assessments will be conducted for all groups at baseline (T1), thereafter the intervention groups will undergo a 5-weeks 15-hour ARTISAN intergenerational arts programme that integrates curated museum visits, facilitated storytelling, creative art-making, and reflective writing for exploring and sharing life narratives on heritage, adversity, strengths and unity, with the aim to foster aspirations, resilience, wellbeing and social cohesion. Upon completion of programme among the intervention group, all 4 groups will be assessed again (T2), and thereafter, the wait-listed controlled group will received the same 5-week 15-hour programme. At the end of all intervention components, a final exit assessment will be conducted on all groups (T3).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Youths and seniors in the intervention group will be paired to receive a novel five-week (3 hours/ week) bilingual (English/ Mandarin), intergenerational arts programme which includes guided museum tours, collaborative art-making and story telling as well as reflective writing. These sessions will be held at the National Museum, and facilitated by experienced artists and trained art therapists.
  Interventions: Behavioral: ARTISAN
- Waitlist Control Group (Experimental): Participants will serve as a waitlist control group before receiving the intervention that the intervention group receives at the end of 5 weeks.
  Interventions: Behavioral: ARTISAN

INTERVENTIONS:
Behavioral: ARTISAN — In the first four weeks, dyads will engage in museum tours facilitated by a docent from the National Museum, followed by a guided storytelling/art-making session (inspired by the artifacts in the gallery), writing activity and group sharing/debrief. The first three weeks of art making will be pair-work by the seniors and youth, while the fourth week will be a collaborative art piece that is created by all participants in the working group. In the last week, the participants will be involved in a mini-exhibition where they will share their works with the group and members of the public, and engage in guided reflection on each other's artworks.
  The main content and discussion point for each session are as follows:
  * Week 1: Food and Play as our National Heritage
  * Week 2: Our Voices, Our Singapore: Strengthening Bonds
  * Week 3: Overcoming Adversities: Stories of Resilience
  * Week 4: Beholding the Future: Dreams and Aspirations
  * Week 5: Passing It On: The Stories We Share

SUMMARY:
This pilot study adopts a Participatory Action Research (PAR) approach to develop a novel ARTISAN intergenerational arts programme that aims to promote life meaning, resilience and wellbeing, as well as to enhance social support and national identity, among the older and younger generations Singapore. Utilizing a wait-list Randomized Controlled Trial design, 30 elderlies and 30 youths (N=60) will be invited to participate in a 5-weeks, 10-hours intervention programme.

Through the integrative processes of curated museum visits (art space), facilitated storytelling (art facilitation), creative art-making and reflective writing (art content), the intervention will focus on the exploration of five unique themes to engage senior-youth dyads. They include: (a) Discovering National Heritage, (b) Strengthening Social Bonds, (c) Overcoming Adversities and Resilience, (d) Building Dreams and Aspirations, and (e) Sharing Stories and Legacies.

Quantitative data obtained before and after the intervention will be triangulated with qualitative data generated from feasibility focus groups and reflective writings to explore its potential benefits and benefiting processes in achieving the aforementioned outcomes. To encourage social change and empowerment, public art exhibitions showcasing the artworks from this programme will also be held within the community. The findings from this study will form the foundation for a larger Population Health Project on Arts and Wellness.

DETAILED DESCRIPTION:
Research Objectives

In order to foster and cultivate aspiration and promote resilience in Singapore, stories of life and strength should be discovered and embraced. Through the reflective and expressive strength of arts, this proposed pilot study - Project ARTISAN: fostering Aspiration & Resilience Through Intergenerational Storytelling & Art-based Narratives - aspires to empower both seniors and youths through intergenerational storytelling and art making to achieve the following objectives:

1. Empowerment: This research will develop and evaluate a novel, cultural-specific ARTISAN intergenerational arts programme with the aim to enhance youths' and seniors' sense life meaning, resilience and wellbeing, leading to greater social cohesion and national identity.
2. Engagement: In the ARTISAN exhibition that showcases the creations generated from the study, the investigators aim to engage families and friends of study participants, as well as members of the public in gaining a renewed understanding towards Singaporean youths and seniors.
3. Social change: Through the development of ARTISAN, the investigators aim to create a platform for intergeneration interaction and knowledge exchange, encouraging the cultivation of positive public social dialogue and change.
4. Sustainability: Findings generated from this study will serve as the empirical foundation for a future Population Health study that aspires toward large-scale implementation of Project ARTISAN in greater community, which can in turn benefit more participants from different walks of life.

Methodology

This pilot study adopts a Participatory Action Research (PAR) approach to develop a novel ARTISAN intergenerational arts programme that aims to promote life meaning, resilience and wellbeing, as well as to enhance social support and national identity, among the older and younger generations Singapore. Utilizing a wait-list Randomized Controlled Trial (RCT) design, pre, post, and follow-up data will be collected and analysis to evaluate programme effectiveness in achieving the stated objectives. Finally, a feasibility assessment will be carried out to investigate programme acceptability and suitability for local population. Ethical approval will be obtained from Nanyang Technological University's Institutional Review Board. Informed consent will also be sought from the participants to ensure confidentiality, beneficence and non-maleficence.

Sampling. Two groups of research participants will be involved in this study: (a) 30 community dwelling seniors aged 60 and above; and (b) 30 youths aged 18 - 35.

Procedures. Participants from each age group will be paired up to form one-to-one senior-youth dyads that will remain intact for the full project duration upon successful recruitment and informed consent, each dyads will then be randomized into 4 groups comprising 7-8 dyads each, with 2 intervention groups and 2 wait-list control group. Wellbeing and self-concept assessments will be conducted for all groups at baseline (T1), thereafter the intervention groups will undergo a 5-weeks 15-hour ARTISAN intergenerational arts programme that integrates curated museum visits, facilitated storytelling, creative art-making, and reflective writing for exploring and sharing life narratives on heritage, adversity, strengths and unity, with the aim to foster aspirations, resilience, wellbeing and social cohesion. Upon completion of programme among the intervention group, all 4 groups will be assessed again (T2), and thereafter, the wait-listed controlled group will received the same 5-week 15-hour programme. At the end of all intervention components, a final exit assessment will be conducted on all groups (T3). A public art exhibition will also be held at the end of the programme to reach out to friends and relatives of the participants, as well as the members of the public. If possible, the art pieces will be permanently showcased within the community. During the art exhibition, exhibition viewers will be encouraged to respond and reflect upon the artworks.

To assess the implementation and delivery of the ARTISAN intergenerational arts programme in community settings, time needed to organize and conduct the intervention sessions, deviations from the intervention protocol and uncompleted interventions and the reasons; as well as the programme leaders' perceptions of competence as a result of training, will be recorded. Programme leaders will also record their experiences of delivering the intervention, their observations of participants' responses during and after the intervention, as well as any difficult or deviant cases. Finally, a randomly selected 24 study participants will be invited to participate in 4 feasibility focus groups after completion of the pilot study (2 groups for 12 seniors and 2 groups for 12 youths). The purpose of these focus groups is to explore and elicit the lived experiences of participants going through Project ARTISAN, allowing space for them to share their thoughts, feelings and personal meaning and benefits of the programme, as well as to elicit their views on the inner workings of the programme so as to offer feedbacks for programme enhancement. All focus group sessions will be recorded, transcribed verbatim and analyzed using thematic framework analysis.

Significance and Uniqueness of Research

Project ARTISAN utilizes the methods of participatory action research in identifying the needs, raising the voices, and illuminating the lives of both seniors and youths in Singapore who are increasingly faced with the challenges of social isolation and decreasing mental health. Through an unique integrative approach that examines the interplay between curated art space, art content and art facilitation, it further aspires to develop a structured intervention protocol for enhancing participants' aspirations, resilience, personhood and nationhood, one that can be adopted and implemented widely across all art, education, health and social care settings in the local context. In sum, this first-of-its-kind study fills a critical gap in knowledge and practice between the intersection of arts, health and culture, while fostering community engagement for enhancing societal wellbeing and social cohesion.

ELIGIBILITY:
Inclusion Criteria:

* Youths: Aged 18 to 35
* Seniors: Aged 60 and above
* No mobility issues
* Able to provide informed consent (or assent)
* Not suffering from major mental health problems

Exclusion Criteria:

* Unable to provide consent
* Suffering from major mental health problems

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Ego-Resilience | Participants will be assessed at three time points: [T1] baseline; [T2] immediately post-intervention/second baseline (5 weeks post T1); and [T3] 5 weeks follow-up/ immediately post-intervention (5 weeks post T2)
  The 14-item Ego-Resilience Revised Scale (ER-89) assesses trait resilience. Participants will be asked to indicate their agreement for statements on a 7-point likert scale. Overall average scores and subscale scores on Active engagement with the world, Integrated performance under stress and Repertoire of (social, personal and cognitive) problem solving strategies will be calculated. Higher values represent greater levels of resilience.
Social Connectedness | Participants will be assessed at three time points: [T1] baseline; [T2] immediately post-intervention/second baseline (5 weeks post T1); and [T3] 5 weeks follow-up/ immediately post-intervention (5 weeks post T2)
  The 8-item Social Connectedness Scale (SCS) assesses Social Connectedness. Participants will be asked to indicate their agreement for statements on a 6-point likert scale. An overall score will be calculated, with higher scores reflecting a greater sense of connectedness. Potential scores range from 8 - 48.
National Identity | Participants will be assessed at three time points: [T1] baseline; [T2] immediately post-intervention/second baseline (5 weeks post T1); and [T3] 5 weeks follow-up/ immediately post-intervention (5 weeks post T2)
  The revised 15-item National Identity Scale (NATID) assesses multiple domains of National Identity. Participants will be asked to indicate their agreement for statements on a 7-point likert scale. Overall average subscale scores for National Heritage, Culture Homogeneity and Belief system will be calculated. Higher values represent greater levels of National Identity.
Loneliness | Participants will be assessed at three time points: [T1] baseline; [T2] immediately post-intervention/second baseline (5 weeks post T1); and [T3] 5 weeks follow-up/ immediately post-intervention (5 weeks post T2)
  The 8-item UCLA Loneliness Scale (ULS-8) assesses Loneliness. Participants will be asked to indicate their agreement for statements on a 4-point scale. An overall score will be calculated, with higher scores reflecting a greater sense of loneliness. Potential score ranges from 8 - 32.

SECONDARY OUTCOMES:
Quality of Life | Participants will be assessed at three time points: [T1] baseline; [T2] immediately post-intervention/second baseline (5 weeks post T1); and [T3] 5 weeks follow-up/ immediately post-intervention (5 weeks post T2)
  The 8-item World Health Organization Quality of Life Scale-8 (WHOQoL-8) measures subjective quality of life. Participants will be asked to respond to questions about areas of their lives on a 5-point likert scale. An overall score will be calculated, with higher values representing greater quality of life. Potential scores range from 8 - 40.
Life Satisfaction | Participants will be assessed at three time points: [T1] baseline; [T2] immediately post-intervention/second baseline (5 weeks post T1); and [T3] 5 weeks follow-up/ immediately post-intervention (5 weeks post T2)
  The single-item Satisfaction with Life Scale (SWLS) measures life satisfaction. Participants will be asked to respond on a 4-point scale with higher values representing better life satisfaction.
Life Meaning | Participants will be assessed at three time points: [T1] baseline; [T2] immediately post-intervention/second baseline (5 weeks post T1); and [T3] 5 weeks follow-up/ immediately post-intervention (5 weeks post T2)
  The 'Presence of Meaning' Subscale from the Meaning in Life Questionnaire (MLQ) is a 5-item measure to assess the participant's sense of meaning in life. Participants will be asked to respond to statements about meaning on a 7-point scale with higher scores indicating a greater sense of life meaning. An overall score will be calculated.
Compassion | Participants will be assessed at three time points: [T1] baseline; [T2] immediately post-intervention/second baseline (5 weeks post T1); and [T3] 5 weeks follow-up/ immediately post-intervention (5 weeks post T2)
  The 5-item Santa Clara Brief Compassion Scale (SCBCS) measures participant's sense of compassion towards others. Participants will be asked to rate statements on a 7-point scale. An overall average score will be calculated, with larger values representing a higher degree of compassion.
Social Support | Participants will be assessed at three time points: [T1] baseline; [T2] immediately post-intervention/second baseline (5 weeks post T1); and [T3] 5 weeks follow-up/ immediately post-intervention (5 weeks post T2)
  Three subscales from the Medical Outcomes Study Social Support Survey (MOS-SS) will be used to measure social support. Specifically, the 8-item Emotional/Informational Support subscale, the 4-item Positive Social Interactions as well as the 3-item Affectionate Support. Participants will be asked to rate on a 5-point likert scale. Subscale scores will be calculated, with higher values representing greater sense of social support.

CONTACTS AND LOCATIONS:
Overall Officials: Andy HY Ho, Principal Investigator — Nanyang Techological University
Locations (1):
- Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ho, A.H.Y., Chui, C.H.K., Borschel, M. (2017). Understanding and managing youth and elderly suicide in Developed East Asia: The imperative of compassion in public health. In G. Cox & N. Thompson (eds.), Handbook of Traumatic Loss: A Guild to Theory and Practice (Chapter 8, pp. 107-122). UK: Routledge.
- [Background] Ho, A.H.Y. (2017). The Arts for Ageing Well: A Singapore Experience. Keynote Speaker at the Arts in Eldercare Symposium 2017. Singapore, 6 September 2017.
- [Background] Ho, A.H.Y., Ho, R.H.M., Pang, J. Ortega, E., & Ma, S.H.X. (2018). Research Report on the Arts for Ageing Well - A Landscape Study on Art Participation and Holistic Wellbeing among Current and Future Older Generations of Singapore. Singapore: Action Research for Community Health, Nanyang Technological University.
- [Background] Ho, A.H.Y., & Tan-Ho, G. (2018) Mindful-Compassion Art Therapy: A Handbook for Practitioners. Singapore: Action Research for Community Health (ARCH), Psychology, School of Social Sciences, Nanyang Technological University.
- [Background] Ho, R.T.H., Potash, J.S., Ho, A.H.Y., Ho, V.F.L. & Chen, E.Y.H. (2016). Reducing mental illness stigma and fostering empathic citizenship: Community arts collaborative approach. Social Work in Mental Health, 15(4), 469-485, DOI: 10.1080/15332985.2016.1236767